CLINICAL TRIAL: NCT03232580
Title: Phase II Study of 99mTc-rhAnnexin V-128 Radionuclide Imaging in Patients With Clinical Suspicion or Confirmed Diagnosis of Spondyloarthritis (SpA)
Brief Title: 99mTc-rhAnnexin V-128 in Diagnosis of Spondyloarthritis
Acronym: Annexin 03
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision based on strategic considerations.
Sponsor: Advanced Accelerator Applications (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AAA-Annexin-03; CAAA113A22201 (Other: Novartis)
Record Dates: First submitted 2017-07-13; First posted 2017-07-28 (Actual); Results first posted 2019-12-13 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Spondyloarthritis
Keywords: Suspicion or confirmed diagnosis of Spondyloarthritis; Ankylosing Spondylarthritis; Ankylosing Spondylitis; Ankylosing Spondyloarthritis; Rheumatoid Spondylitis; Spondylarthritis Ankylopoietica; Spondylitis Ankylopoietica; Spondyloarthritis Ankylopoietica; Autoimmune systemic rheumatic disease; Inflammatory bowel disease; Psoriatic arthritis; Undifferentiated spondyloarthropathy.
MeSH Terms: conditions — Spondylarthritis; Spondylitis, Ankylosing; Inflammatory Bowel Diseases; Arthritis, Psoriatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- rhAnnexin V-128 (Experimental): All patients received a single i.v injection of 99mTc-rhAnnexin V-128 at Day 0.
  Interventions: Drug: rhAnnexin V-128

INTERVENTIONS:
Drug: rhAnnexin V-128 — All patients received a single i.v injection of 99mTc-rhAnnexin V-128 at Day 0.

SUMMARY:
This single center, open-label, proof of concept (PoC) Phase II study aimed to assess the investigational imaging agent 99mTc-rhAnnexin V-128 in detecting spondyloarthritis (SpA) lesions.

Overall, it was planned to recruit 20 adults with suspected or confirmed SpA. First, 5 patients were enrolled into a "proof of concept" phase, to assess the imaging potential of 99mTc-rhAnnexin V-128 in terms of imaging quality, disease-lesion radiotracer uptake and medical relevance. Based on these results the Data Monitoring Committee (DMC) was to decide whether to terminate the study or whether to continue and enroll the next 15 planned patients.

DETAILED DESCRIPTION:
The study was prematurely terminated by the sponsor after the first 5 patients completed the PoC phase based on strategic considerations.

Novartis acquired Advanced Accelerator Applications SA.

ELIGIBILITY:
Inclusion Criteria:

For the first 5 patients enrolled in the POC part:

1. Patients with clinical suspicion or confirmed diagnosis of SpA, based on the ASA criteria with active symptoms including back, hip or buttock pain prior to:

* A change in NSAID therapy or
* A change in non-biologic DMARD or
* A start of non-biologic DMARD.

For the next 15 patients enrolled in the Phase II part:

1. Patients with clinical suspicion or confirmed diagnosis of SpA, based on the ASAS criteria with active symptoms including back, hip or buttock pain prior to:

   * A change in NSAIDs therapy
   * A change in non-biologic DMARD
   * A start of non-biologic DMARD
   * A start of biologic DMARD

   For all patients:
2. Age over 18 years old.
3. Signed Informed Consent Form

Exclusion Criteria:

1. Pregnancy or lactation
2. Liver impairment (ALT, AST or Bilirubin > 2 ULN) at screening visit or baseline
3. Kidney impairment (serum creatinine > 1.5 mg/dL)
4. History of any disease or relevant physical or psychiatric condition or abnormal physical finding which may interfere with the study objectives at the investigator judgment
5. Known hypersensitivity to the investigational drug or any of its components
6. Contraindication(s) to the MRI procedure (claustrophobia, prosthetic valve, pacemaker, inability to lie still in a supine position)
7. Participation to another clinical trial within 4 weeks before study inclusion except for patients who have participated or who are currently participating in an interventional study without any study drug administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2018-11-12 (Actual); Study Completion 2018-11-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 5 patients enrolled single site in US
Period: Overall Study
Arm/Group | rhAnnexin V-128
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | rhAnnexin V-128
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 4
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic | 2
  Caucasian | 3
Participants with Magnetic Resonance Imaging (MRI) results at Screening [Count of Participants; unit: Participants] — All patients had a routine MRI to assess SpA induced inflammation in the sacroiliac and lumbar spine joints.
  Participants
    MRI Results in Lumbar Spine: Negative | 4
    MRI Results in Lumbar Spine: Positive | 1
    MRI Results in Sacroiliac Joints: Negative | 4
    MRI Results in Sacroiliac Joints: Positive | 1
Participants with Clinical Pain at Screening [Count of Participants; unit: Participants]
  Clinical Pain in Lumbar Spine: Yes | 5
  Clinical Pain in Lumbar Spine: No | 0
  Clinical Pain in Sacroiliac Joints: Yes | 5
  Clinical Pain in Sacroiliac Joints: No | 0

OUTCOME MEASURES:

1. Primary Outcome: 99mTc-rhAnnexin V-128 Uptake
Description: In order to asses 99mTc-rhAnnexin V-128 magnitude and dynamic range of uptake within areas affected by inflammation, Single-Photon Emission Computed Tomography (SPECT)/Computed Tomography (CT) scans were interpreted and graded by at least two independent experienced nuclear medicine physicians blinded from clinical data and other imagings modality results.
  Uptake compared with background (e.g. physiological liver uptake) were assessed for each affected area by nuclear medicine physicians using a 4-grade scoring system (e.g. 0, none; 1, mild or present but < to background uptake; 2, moderate or = to background uptake; 3, intense or > to background uptake). Only descriptive analysis performed.
Time Frame: 60 minutes and 120 minutes post investigational product adminstration
Population: Only participants with a grading uptake at any given body region are included in the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | rhAnnexin V-128
Number analyzed (Participants) | 5
Participants
  60 minutes: Whole Body Planar - Principal Inv.: Grade of uptake = 0 | 2
  60 minutes: Whole Body Planar - Principal Inv.: Grade of uptake = 1 | 1
  60 minutes: Whole Body Planar - Principal Inv.: Grade of uptake = 2 | 2
  60 minutes: Whole Body Planar - Principal Inv.: Grade of uptake = 3 | 0
  60 minutes: Whole Body Planar - Reviewer 1: Grade of uptake = 0 | 5
  60 minutes: Whole Body Planar - Reviewer 1: Grade of uptake = 1 | 0
  60 minutes: Whole Body Planar - Reviewer 1: Grade of uptake = 2 | 0
  60 minutes: Whole Body Planar - Reviewer 1: Grade of uptake = 3 | 0
  60 minutes: Whole Body Planar - Reviewer 2: Grade of uptake = 0 | 3
  60 minutes: Whole Body Planar - Reviewer 2: Grade of uptake = 1 | 2
  60 minutes: Whole Body Planar - Reviewer 2: Grade of uptake = 2 | 0
  60 minutes: Whole Body Planar - Reviewer 2: Grade of uptake = 3 | 0
  120 minutes: Whole Body Planar - Principal Inv.: number analyzed (Participants) | 4
  120 minutes: Whole Body Planar - Principal Inv.: Grade of uptake = 0 | 1
  120 minutes: Whole Body Planar - Principal Inv.: Grade of uptake = 1 | 2
  120 minutes: Whole Body Planar - Principal Inv.: Grade of uptake = 2 | 1
  120 minutes: Whole Body Planar - Principal Inv.: Grade of uptake = 3 | 0
  120 minutes: Whole Body Planar - Reviewer 1: Grade of uptake = 0 | 5
  120 minutes: Whole Body Planar - Reviewer 1: Grade of uptake = 1 | 0
  120 minutes: Whole Body Planar - Reviewer 1: Grade of uptake = 2 | 0
  120 minutes: Whole Body Planar - Reviewer 1: Grade of uptake = 3 | 0
  120 minutes: Whole Body Planar - Reviewer 2: Grade of uptake = 0 | 3
  120 minutes: Whole Body Planar - Reviewer 2: Grade of uptake = 1 | 2
  120 minutes: Whole Body Planar - Reviewer 2: Grade of uptake = 2 | 0
  120 minutes: Whole Body Planar - Reviewer 2: Grade of uptake = 3 | 0
  60 minutes: Abdomen - Principal Inv.: Grade of uptake = 0 | 4
  60 minutes: Abdomen - Principal Inv.: Grade of uptake = 1 | 1
  60 minutes: Abdomen - Principal Inv.: Grade of uptake = 2 | 0
  60 minutes: Abdomen - Principal Inv.: Grade of uptake = 3 | 0
  60 minutes: Abdomen - Reviewer 1: Grade of uptake = 0 | 5
  60 minutes: Abdomen - Reviewer 1: Grade of uptake = 1 | 0
  60 minutes: Abdomen - Reviewer 1: Grade of uptake = 2 | 0
  60 minutes: Abdomen - Reviewer 1: Grade of uptake = 3 | 0
  60 minutes: Abdomen - Reviewer 2: Grade of uptake = 0 | 5
  60 minutes: Abdomen - Reviewer 2: Grade of uptake = 1 | 0
  60 minutes: Abdomen - Reviewer 2: Grade of uptake = 2 | 0
  60 minutes: Abdomen - Reviewer 2: Grade of uptake = 3 | 0
  120 minutes: Abdomen - Principal Inv.: Grade of uptake = 0 | 4
  120 minutes: Abdomen - Principal Inv.: Grade of uptake = 1 | 0
  120 minutes: Abdomen - Principal Inv.: Grade of uptake = 2 | 1
  120 minutes: Abdomen - Principal Inv.: Grade of uptake = 3 | 0
  120 minutes: Abdomen - Reviewer 1: Grade of uptake = 0 | 5
  120 minutes: Abdomen - Reviewer 1: Grade of uptake = 1 | 0
  120 minutes: Abdomen - Reviewer 1: Grade of uptake = 2 | 0
  120 minutes: Abdomen - Reviewer 1: Grade of uptake = 3 | 0
  120 minutes: Abdomen - Reviewer 2: Grade of uptake = 0 | 5
  120 minutes: Abdomen - Reviewer 2: Grade of uptake = 1 | 0
  120 minutes: Abdomen - Reviewer 2: Grade of uptake = 2 | 0
  120 minutes: Abdomen - Reviewer 2: Grade of uptake = 3 | 0
  60 minutes: Lumbosacral - Principal Inv.: Grade of uptake = 0 | 2
  60 minutes: Lumbosacral - Principal Inv.: Grade of uptake = 1 | 0
  60 minutes: Lumbosacral - Principal Inv.: Grade of uptake = 2 | 3
  60 minutes: Lumbosacral - Principal Inv.: Grade of uptake = 3 | 0
  60 minutes: Lumbosacral - Reviewer 1: Grade of uptake = 0 | 3
  60 minutes: Lumbosacral - Reviewer 1: Grade of uptake = 1 | 2
  60 minutes: Lumbosacral - Reviewer 1: Grade of uptake = 2 | 0
  60 minutes: Lumbosacral - Reviewer 1: Grade of uptake = 3 | 0
  60 minutes: Lumbosacral - Reviewer 2: Grade of uptake = 0 | 5
  60 minutes: Lumbosacral - Reviewer 2: Grade of uptake = 1 | 0
  60 minutes: Lumbosacral - Reviewer 2: Grade of uptake = 2 | 0
  60 minutes: Lumbosacral - Reviewer 2: Grade of uptake = 3 | 0
  120 minutes: Lumbosacral - Principal Inv.: number analyzed (Participants) | 4
  120 minutes: Lumbosacral - Principal Inv.: Grade of uptake = 0 | 2
  120 minutes: Lumbosacral - Principal Inv.: Grade of uptake = 1 | 0
  120 minutes: Lumbosacral - Principal Inv.: Grade of uptake = 2 | 2
  120 minutes: Lumbosacral - Principal Inv.: Grade of uptake = 3 | 0
  120 minutes: Lumbosacral - Reviewer 1: Grade of uptake = 0 | 3
  120 minutes: Lumbosacral - Reviewer 1: Grade of uptake = 1 | 2
  120 minutes: Lumbosacral - Reviewer 1: Grade of uptake = 2 | 0
  120 minutes: Lumbosacral - Reviewer 1: Grade of uptake = 3 | 0
  120 minutes: Lumbosacral - Reviewer 2: Grade of uptake = 0 | 5
  120 minutes: Lumbosacral - Reviewer 2: Grade of uptake = 1 | 0
  120 minutes: Lumbosacral - Reviewer 2: Grade of uptake = 2 | 0
  120 minutes: Lumbosacral - Reviewer 2: Grade of uptake = 3 | 0
  60 minutes: Sacroiliac Joint - Principal Inv.: Grade of uptake = 0 | 2
  60 minutes: Sacroiliac Joint - Principal Inv.: Grade of uptake = 1 | 0
  60 minutes: Sacroiliac Joint - Principal Inv.: Grade of uptake = 2 | 3
  60 minutes: Sacroiliac Joint - Principal Inv.: Grade of uptake = 3 | 0
  60 minutes: Sacroiliac Joint - Reviewer 1: Grade of uptake = 0 | 5
  60 minutes: Sacroiliac Joint - Reviewer 1: Grade of uptake = 1 | 0
  60 minutes: Sacroiliac Joint - Reviewer 1: Grade of uptake = 2 | 0
  60 minutes: Sacroiliac Joint - Reviewer 1: Grade of uptake = 3 | 0
  60 minutes: Sacroiliac Joint - Reviewer 2: Grade of uptake = 0 | 4
  60 minutes: Sacroiliac Joint - Reviewer 2: Grade of uptake = 1 | 1
  60 minutes: Sacroiliac Joint - Reviewer 2: Grade of uptake = 2 | 0
  60 minutes: Sacroiliac Joint - Reviewer 2: Grade of uptake = 3 | 0
  120 minutes: Sacroiliac Joint - Principal Inv.: number analyzed (Participants) | 4
  120 minutes: Sacroiliac Joint - Principal Inv.: Grade of uptake = 0 | 1
  120 minutes: Sacroiliac Joint - Principal Inv.: Grade of uptake = 1 | 1
  120 minutes: Sacroiliac Joint - Principal Inv.: Grade of uptake = 2 | 2
  120 minutes: Sacroiliac Joint - Principal Inv.: Grade of uptake = 3 | 0
  120 minutes: Sacroiliac Joint - Reviewer 1: Grade of uptake = 0 | 5
  120 minutes: Sacroiliac Joint - Reviewer 1: Grade of uptake = 1 | 0
  120 minutes: Sacroiliac Joint - Reviewer 1: Grade of uptake = 2 | 0
  120 minutes: Sacroiliac Joint - Reviewer 1: Grade of uptake = 3 | 0
  120 minutes: Sacroiliac Joint - Reviewer 2: Grade of uptake = 0 | 4
  120 minutes: Sacroiliac Joint - Reviewer 2: Grade of uptake = 1 | 1
  120 minutes: Sacroiliac Joint - Reviewer 2: Grade of uptake = 2 | 0
  120 minutes: Sacroiliac Joint - Reviewer 2: Grade of uptake = 3 | 0

2. Primary Outcome: 99mTc-rhAnnexin V-128 Uptake Adjudication
Description: In order to asses 99mTc-rhAnnexin V-128 magnitude and dynamic range of uptake within areas affected by inflammation, Single-Photon Emission Computed Tomography (SPECT)/Computed Tomography (CT) scans were interpreted and graded by at least two independent experienced nuclear medicine physicians blinded from clinical data and other imagings modality results.
  In case of discrepancies between the different readers, an adjudication process based on consensus was put in place in order to obtain one final outcome for each area. Adjudication results were categorized as Positive or Negative. Only descriptive analysis performed.
Time Frame: 60 minutes and 120 minutes post investigational product adminstration
Measure: Count of Participants; unit: Participants
Arm/Group | rhAnnexin V-128
Number analyzed (Participants) | 5
Participants
  Whole Body Planar - 60 minutes: Positive | 1
  Whole Body Planar - 60 minutes: Negative | 4
  Whole Body Planar - 120 minutes: Positive | 2
  Whole Body Planar - 120 minutes: Negative | 3
  Abdomen - 60 minutes: Positive | 0
  Abdomen - 60 minutes: Negative | 5
  Abdomen - 120 minutes: Positive | 0
  Abdomen - 120 minutes: Negative | 5
  Lumbosacral - 60 minutes: Positive | 2
  Lumbosacral - 60 minutes: Negative | 3
  Lumbosacral - 120 minutes: Positive | 2
  Lumbosacral - 120 minutes: Negative | 3
  Sacroiliac - 60 minutes: Positive | 1
  Sacroiliac - 60 minutes: Negative | 4
  Sacroiliac - 120 minutes: Positive | 1
  Sacroiliac - 120 minutes: Negative | 4

ADVERSE EVENTS:
Time Frame: Adverse event were collected from first dosing (single administration, Day 0) plus 30 days post-treatment.
Description: Any signs or symptom that occurs during the study treatment plus 30 days post-treatment.
Arm/Group | rhAnnexin V-128
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 2/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rhAnnexin V-128 (N=5)
Nausea (Injury, poisoning and procedural complications) | 1 (1)
Itching at injection site (Injury, poisoning and procedural complications) | 1 (1)
Redness at injection site (Injury, poisoning and procedural complications) | 1 (1)
Head cold (Respiratory, thoracic and mediastinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
After the first 5 patients completed the Proof of Concept (PoC) phase, the study was terminated based on strategic considerations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-03-13): https://cdn.clinicaltrials.gov/large-docs/80/NCT03232580/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-06): https://cdn.clinicaltrials.gov/large-docs/80/NCT03232580/SAP_001.pdf